CLINICAL TRIAL: NCT04474457
Title: An ObservationaI Study to Evaluate the Efficacy and Safety of Favipiravir in the Treatment of COVID-19 Patients Over 15 Years of Age Who Are Receiving Favipiravir
Brief Title: Efficacy and Safety of Favipiravir in the Treatment of COVID-19 Patients Over 15 Years of Age
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ministry of Health, Turkey (Other Government)
Collaborators: Hacettepe University (Other); Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other); Umraniye Education and Research Hospital (Other Government); Istanbul Training and Research Hospital (Other Government); Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other); Tepecik Training and Research Hospital (Other); Istanbul University - Cerrahpasa (Other); Ankara University (Other); Ankara City Hospital Bilkent (Other); Ankara Training and Research Hospital (Other); Ege University Hospital (Application and Research Center) (Unknown); Derince Training and Research Hospital (Other); Istanbul University (Other); Kayseri City Hospital (Other Government)
Responsible Party: Principal Investigator, Prof. Ates KARA, MD, Prof., Hacettepe University
Other Study IDs: COVID-19-PMS-FAV
Record Dates: First submitted 2020-07-15; First posted 2020-07-16 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — favipiravir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19/Favipiravir: Turkish patient cohort diagnosed with COVID-19 and previously initiated treatment with "Favipiravir".
  Interventions: Drug: Favipiravir

INTERVENTIONS:
Drug: Favipiravir — Turkish patient cohort diagnosed with COVID-19 and previously initiated treatment with "Favipiravir".

SUMMARY:
This study is an observational study (Non-interventional study) to evaluate the safety and efficacy of favipiravir in patients older than 15 years of age, diagnosed with COVID-19 and initiated treatment with favipiravir before enrollment to the study. Patients who have already had a routine favipiravir treatment decision or alternatively favipiravir treatment started at the time of enrollment, will be included in this study.

DETAILED DESCRIPTION:
The clinical picture of 2019-nCoV disease is in a broad spectrum, which includes asymptomatic infection, a mild upper respiratory tract infection, respiratory failure, and even severe viral pneumonia with death. Although the mortality rate is not yet clear, the reported case-fatality risk was 11-14% during the initial studies which included patients with severe disease. The overall case fatality rate was reported as approximately 2%. In addition, most cases have resulted in a pneumonia requiring supplemental oxygen therapy and ventilator support. The alarming levels of spread and severity of COVID-19 caused a global emergency and this outbreak has been characterized as a pandemic by the World Health Organization (WHO).

Studies have suggested that investigational product favipiravir can improve the recovery of patients with mild disease and reduce the treatment duration from less than 11 days.

The main purpose of this study is to obtain efficacy and safety data for favipiravir use in the Turkish patient cohort diagnosed with COVID-19 and decided to be treated with "Favipiravir" before enrollment to this observational study. This study is designed as an observational drug study which will evaluate the safety and efficacy of favipiravir in patients and diagnosed with COVID-19 and older than 15 years of age.

This study is designed as an observational drug study to evaluate the safety and efficacy of favipiravir in patients diagnosed with COVID-19 and older than 15 years of age with a favipiravir treatment decision. Patients who have already had a routine favipiravir treatment decision or favipiravir treatment started will be included in this study.

A total of 1000 female and male patients aged 15 years or older will be included in the study. The planned observation duration for each patient is 7 days.

This study will be conducted in 14 sites.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, diagnosed with Covid-19 disease who are 15 years of age or older at the time of enrollment
* Patients who have understood all study procedures that will be applied under the study protocol
* Patients with confirmed diagnosis of COVID-19 by PCR and/or other accepted methods and have a treatment decision with favipiravir
* Patients who will accept oropharyngeal sample and venous blood sample collection periodically within the scope of the study protocol

Exclusion Criteria:

* Patients who are pregnant or females who are breast feeding
* Patients under the age of 15

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1000 patients aged 15 years or older and diagnosed with COVID-19 who meet inclusion/exclusion criteria of the study and have decision of treatment with favipiravir .
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Time to recovery (discharge) | 7 days
  The evaluation of the recovery discharge until the 7th day of hospitalization after the initiation of treatment.
Decrease in viral load | 7 days
  The evaluation of decrease in viral load until 7th day hospitalization after the initiation of treatment.

SECONDARY OUTCOMES:
Adverse Event (AE), Serious Adverse Event (SAE) and discontinuation of treatment | 7 days
  Number/characteristics of Adverse Event (AE), Serious Adverse Event (SAE) and discontinuation of treatment due to study drug from baseline until the end of study.
Frequency of occurrence of lymphopenia from baseline | 7 days
  Clinical evaluation of occurrence of lymphopenia from baseline until the end of study.
Frequency of occurrence of thrombocytopenia from baseline | 7 days
  Clinical evaluation of occurrence of thrombocytopenia from baseline until the end of study.
Changes in alanine aminotransferase (ALT) levels from baseline | 7 days
  Clinical evaluation of ALT levels from baseline until the end of study.
Changes in aspartate aminotransferase (AST) levels from baseline | 7 days
  Clinical evaluation of AST levels from baseline until the end of study.
Changes in C-reactive protein (CRP) levels from baseline | 7 days
  Clinical evaluation of CRP levels from baseline until the end of study.
Changes in level of D-dimer levels from baseline | 7 days
  Clinical evaluation of D-dimer levels from baseline until the end of study.
Changes in prothrombin time (PT) values from baseline | 7 days
  Clinical evaluation of PT values for blood to coagulate from baseline until the end of study.
Changes in partial thromboplastin time (PTT) values from baseline | 7 days
  Clinical evaluation of PTT values for blood to coagulate from baseline until the end of study.
Changes in blood pressure from baseline | 7 days
  Clinical evaluation of systolic and diastolic blood pressure levels from baseline until the end of study.
Changes in respiratory rate from baseline | 7 days
  Clinical evaluation of respiratory rate levels from baseline until the end of study.
Changes in pulse oximetry from baseline | 7 days
  Clinical evaluation of pulse oximetry levels from baseline until the end of study.
Changes in fever from baseline | 7 days
  Clinical evaluation of changes in fever from baseline until the end of study.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, School of Medicine, Ankara, Turkey (Türkiye)